CLINICAL TRIAL: NCT03003806
Title: Evaluation of the Dreamed Advisor Pro for Automated Insulin Pump Setting Adjustments in Children and Adolescents With Type 1 Diabetes- Open Label, Parallel , Randomized, Controlled Multicenter Study-The Advice4U Pro Study
Brief Title: Evaluation of the Dreamed Advisor Pro for Automated Insulin Pump Setting Adjustments in Children and Adolescents With Type 1 Diabetes- The Advice4U Pro Study
Acronym: Advice4U
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: DreaMed (Industry); The Leona M. and Harry B. Helmsley Charitable Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC072016ctil
Record Dates: First submitted 2016-12-22; First posted 2016-12-28 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2019-06

CONDITIONS: Type1 Diabetes Mellitus
Keywords: Insulin pump treatment; Type 1 diabetes; Pump setting advisor
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DreaMed Advisor Pro (Experimental): Insulin pump settings (i.e, basal plan, correction factor, carbohydrate ratio and insulin activity time) will be adjusted using the DreaMed Advisor Pro
  Interventions: Device: DreaMed Advisor Pro
- Control group-medical guided recommendations (Active Comparator): Insulin pump settings (i.e, basal plan, correction factor, carbohydrate ratio and insulin activity time) will be adjusted by the medical team
  Interventions: Other: Medical guided recommendation

INTERVENTIONS:
Device: DreaMed Advisor Pro — Insulin pump settings (i.e, basal plan, correction factor, carbohydrate ratio and insulin activity time) will be adjusted using the DreaMed Advisor Pro
  Arms: DreaMed Advisor Pro
Other: Medical guided recommendation — Insulin pump settings (i.e, basal plan, correction factor, carbohydrate ratio and insulin activity time) will be adjusted by the medical team
  Arms: Control group-medical guided recommendations

SUMMARY:
The DreaMed Advisor Pro is a software which automatically analyses treatment information, learns patient's needs and accordingly suggests adjustments in insulin dosing. The DreaMed Advisor Pro uses information gathered from glucose monitoring (sensor readings or capillary blood glucose measurements), insulin dosing and meal data during daily routine home care. Following a 5-minute data collection and analysis, the algorithm learns and suggests pump-setting changes for optimization of glucose control

The algorithm is designed as an advisory tool and has three main components:

1. A statistical analysis of the insulin pump and sensor data: insulin delivery, bolus-calculator rate of use, sensor glucose variables, hypoglycemic and hyperglycemia patterns.
2. Practical recommendations, alert messages based on aforementioned data
3. Recommendation for new insulin pump settings: including basal intervals and rate, different carbohydrate ratio according to time of day, correction factor and insulin sensitivity time.

The main goal of the DreaMed Advisor Pro is to improve diabetes management for subjects with Type 1 Diabetes (T1D) by using an innovative Advisor to determine insulin dosing for pump users.

The main objective of the proposed study is to evaluate the safety and efficacy of using the DreaMed Advisor Pro algorithm versus medical guided recommendation to determine insulin dosing for sub-optimal controlled subjects with type 1 diabetes using pump therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject with Type 1 diabetes (>1yr since diagnosis)
* Age ≥ 10 years up to 21 years
* HbA1c at inclusion ≥ 7.0% and ≤ 10%
* Insulin infusion pump therapy: "OmniPod®" Insulin pump (insulet Corp., Bedford, "MA", USA) or any Medtronic pump that is comparable with Glooko app for at least 4 months
* BMI Standard Deviation Score (SDS) - below the 97th percentile for age
* Patients willing to follow study instructions (at least 2 capillary blood glucose readings/day, use the bolus-calculator feature of the pump)
* Patient/ parents are required to have minimum computer skills and understanding of navigating the internet
* Patients willing to use dexcom sensor for the study duration
* Patients/ parents will have to have a smart phone (Apple, Android, Windows)

Exclusion Criteria:

* An episode of diabetic ketoacidosis within the month prior to study entry
* Concomitant diseases/ treatment that influence metabolic control
* Any significant diseases /conditions including psychiatric disorders and substance abuse that in the opinion of the investigator is likely to affect the subject's ability to complete the study or compromise patient's safety,
* Participation in any other interventional study
* Known or suspected allergy to trial products such as adhesives, tapes, needles. An allergy to contrast medium, use of other active medical devices (such as pacemaker, ICD) and planned imaging examinations (such as MRI).
* Female subject who is pregnant or lactating planning to become pregnant within the planned study duration -Severe hypoglycemia six month prior to enrollment as defined by the American Diabetes Association (ADA) and Endocrine Society as follows: "Severe hypoglycemia is an event requiring assistance of another person to actively administer carbohydrates, glucagon, or take other corrective actions". -
* Current use of the following medications: medications that are used to lower blood glucose such as Pramlintide, Metformin and GLP-1 analogs. Beta blockers, glucocorticoids and other medications, which in the judgment of the investigator would be a contraindication to participation in the study (Anticoagulant therapy e.g. Plavix, LMW heparin, Coumadin, Immunosuppressant therapy)
* Relevant severe organ disorders (diabetic nephropathy, diabetic retinopathy, diabetic foot syndrome) or any secondary disease or complication of diabetes mellitus

  * Subject has unstable or rapidly progressive renal disease or is receiving dialysis
  * Subject has active proliferating retinopathy
  * Active gastroparesis
* Patient suffers from an eating disorder

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 122 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
Percentage of glucose readings within range of 70-180 mg/dl (3.9 to 10 mmol/l). | Final visit (week 31)
Percentage of glucose readings below 54 mg/dl (3.3 mmol/l) | Final visit (week 31)

SECONDARY OUTCOMES:
HbA1c | Final visit (week 31)
Percentage of glucose readings below 70 mg/dl (3.9 mmol/L) | Final visit (week 31)
Percentage of readings below 50 mg/dl (2.8 mmol/L) | Final visit (week 31)
Percentage of readings above 180 mg/dl (10.0 mmol/L) | Final visit (week 31)
Percentage of readings above 240 mg/dl (13.3 mmol/L) | Final visit (week 31)
Area above the curve of glucose glucose level of 180 mg/dl | Final visit (week 31)
Area under the curve of glucose level of 70 mg/dl | Final visit (week 31)
Mean sensor blood glucose | Final visit (week 31)
Glucose variability measured by Standard Deviation | Final visit (week 31)
Number of recommendations for changes in settings per patient | Final visit (week 31)
Number of recommendations for changes in settings per iteration | Final visit (week 31)
Number of physician override Advisor recommendations | Final visit (week 31)
Number of patients overrides of recommendation | Final visit (week 31)
Estimated time duration needed for the physician to give its recommendations | Final visit (week 31)
Device satisfaction questionaire | Final visit (week 31)
Diabetes treatment satisfaction questionnaire | Final visit (week 31)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (4):
  - Barbara Davis Center for Childhood Diabetes, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida College of Medicine, Gainesville, Florida
  - Joslin Diabetes Center, One Joslin Place, Boston, Massachusetts
- Diabetes -Zentrum fuer kinder und jugendliche, Hanover, Germany
- Schnider children's medical center, Petah Tikva, Israel
- University Children's Hospital, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nimri R, Battelino T, Laffel LM, Slover RH, Schatz D, Weinzimer SA, Dovc K, Danne T, Phillip M; NextDREAM Consortium. Insulin dose optimization using an automated artificial intelligence-based decision support system in youths with type 1 diabetes. Nat Med. 2020 Sep;26(9):1380-1384. doi: 10.1038/s41591-020-1045-7. Epub 2020 Sep 9. PMID 32908282